CLINICAL TRIAL: NCT04747353
Title: Computed Tomography Targets for Efficient Guidance of Catheter Ablation in Ventricular Tachycardia (MAP-IN-HEART)
Acronym: MAP-IN-HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2021/01
Record Dates: First submitted 2021-01-26; First posted 2021-02-10 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Ventricular Tachycardia
Keywords: Myocardial infarction; Ventricular Tachycardia; Catheter Ablation; Imaging; Cardiac computed tomography
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Catheter ablation procedure performed as part of standard care, although with the addition of an image-based 3D heart model including detailed anatomy and primary ablation targets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catheter ablation procedure with heart 3D model (Experimental): Experimental: Catheter ablation procedure performed as part of standard care, although with the addition of an image-based 3D heart model including detailed anatomy and primary ablation targets
  Interventions: Device: Catheter ablation procedure with heart 3D model

INTERVENTIONS:
Device: Catheter ablation procedure with heart 3D model — Device: Catheter ablation procedure performed as part of standard care, although with the addition of an image-based 3D heart model including detailed anatomy and primary ablation targets

SUMMARY:
The hypothesis of MAP IN HEART is that catheter ablation for post-infarction ventricular tachycardia (VT) can be largely improved through a direct definition of primary ablation targets from pre-operative CT scan imaging. The objective of is to demonstrate that catheter ablation of post-infarction VT targeting left ventricular wall thickness channels as defined from CT scan is feasible and associated with favorable efficacy, efficiency and safety profiles. A single-arm prospective cohort study will be conducted, including 40 patients over 3 European centres. Baseline, procedural and 6-month follow-up data will be analyzed

DETAILED DESCRIPTION:
Background: Although catheter ablation is a recommended therapeutic option in patients with history of myocardial infarction presenting with sustained ventricular tachycardia (VT),1 the current approach relies on lengthy, poorly reproducible and poorly standardized identification of targets derived from invasive catheter measurements. As a consequence, the rate of VT recurrence remains high, leading to repeat interventions.2 Pre-operative CT scan imaging was shown able to identify arrhythmogenic sites within scar through a detailed analysis of left ventricular (LV) wall thickness.3,4 This study aims at demonstrating that using these as primary targets for ablation is a feasible strategy associated with favorable efficacy, efficiency and safety profiles.

Methods: 40 patients with post-infarction VT referred for catheter ablation will be included over 3 European centres. Pre-operative CT scan will be processed to obtain a 3D model of the patient heart comprising detailed anatomy and LV wall thickness maps. Channels of relatively preserved thickness penetrating within severely thinned scar (i.e. CT-channels) will be identified using a proprietary algorithm developed at the IHU LIRYC, University of Bordeaux, and used as primary targets for catheter ablation. During the intervention, the 3D model along with pre-operatively defined targets will be registered in the 3D mapping space, and each CT-channel will be transected by ablation. The inducibility of VT will then be tested and any VT remaining inducible after CT-channels ablation will be targeted using conventional catheter mapping techniques, with a composite procedural endpoint combining the ablation of all CT channels and the non-inducibility of any VT. Procedural and 6-month follow-up data will be analyzed to assess the feasibility of the approach and report its efficiency, efficacy and safety profiles.

Expected results: the CT-guided ablation strategy is expected to be feasible in a vast majority of post-infarction patients referred for VT ablation, and to be extremely time-efficient, the lengthy diagnostic part of the procedure (catheter mapping) being moved pre-operatively (imaging). The short procedure duration should translate into a favorable safety profile. The strategy should also be associated with a high efficacy in eliminating the arrhythmia, thanks to a more comprehensive definition of targets and to the dedication of the procedure time almost entirely to therapy. In conclusion, the present study should provide solid proof of concept on which randomized controlled trials may be built.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for catheter ablation intervention with planned preoperative cardiac CT scan
* Prior myocardial infarction (using the international definition of MI: Q waves or imaging evidence of regional myocardial akinesis/thinning in the absence of a non- ischemic cause with documentation of prior ischemic injury)

and

* One of the following monomorphic VT events within last 6 months:

  * A: ≥3 episodes of symptomatic VT treated with antitachycardia pacing (ATP),
  * B: ≥1 appropriate ICD shocks,
  * C: ≥3 VT episodes within 24 hr
  * D: sustained VT below detection rate of the ICD documented by ECG or any cardiac monitor
  * E: Sustained VT recorded on 12 leads ECG in the absence of ICD
* Signed informed consent
* Affiliated or beneficiary of health insurance

Exclusion Criteria:

* Unable or unwilling to provide written informed consent.
* Active ischemia (acute thrombus diagnosed by coronary angiography, or dynamic ST segment changes demonstrated on ECG) or another reversible cause of VT (e.g. drug-induced arrhythmia), had recent acute coronary syndrome within 30 days thought to be due to acute coronary arterial thrombosis, or have CCS functional class IV angina. Note that biomarker level elevation alone after ventricular arrhythmias does not denote acute coronary syndrome or active ischemia.
* Are known to have protruding left ventricular thrombus or mechanical aortic and mitral valves.
* Have had a prior catheter ablation procedure for VT
* Presenting arrhythmia: polymorphic VT or ventricular fibrillation (VF).
* Are in renal failure (Creatinine clearance <30 mL/min), have NYHA Functional class IV heart failure, or a systemic illness likely to limit survival to <1 year.
* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control. (French HAS criteria or following methods are considered adequate):

  * Combined hormonal contraception
  * Injected hormonal contraception
  * Implanted hormonal contraception
  * Progesterone-only hormonal contraception associated with inhibition of ovulation
  * Placement of an intrauterine device (IUD)
  * Placement of intrauterine hormone-realising system (IUS)
* Patient under legal protection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
evaluation of image-guided VT ablation protocol | end of catheter ablation procedure (hour 3)
  Feasibility of the image-guided VT ablation protocol, defined by the presence of all following criteria:
  * CT imaging acquisition completed (yes/no)
  * pseudonymized images transferred to core lab (yes/no)
  * image processing/3D modeling completed by corelab (yes/no)
  * 3D model transferred to site within 24h of image acquisition (yes/no)
  * 3D model registered in the 3D mapping system during catheter ablation procedure (yes/no)
  * all CT-channels targeted by radiofrequency ablation, regardless of local and procedural outcomes (yes/no)

SECONDARY OUTCOMES:
Rate of acute success after CT-channels ablation | end of catheter ablation procedure (hour 3)
  Rate of acute success after CT-channels ablation, defined as non-inducibility of any VT using a prescribed programmed ventricular stimulation protocol.
Number of VTs persisting after CT channel ablation | end of catheter ablation procedure (hour 3)
  Number of VTs persisting after CT channel ablation
Cycle lengths of VTs persisting after CT channel ablation | end of catheter ablation procedure (hour 3)
  Cycle lengths of VTs persisting after CT channel ablation (ms)
Location of VTs persisting after CT channel ablation | end of catheter ablation procedure (hour 3)
  Location of VTs persisting after CT channel ablation with respect to CT channels. Location (critical isthmuses) will be identified using conventional pace mapping or VT/entrainment mapping methods, and described as matching or not matching the location of one CT channel (yes/no/NA)
Rate of acute success at the end of the procedure | end of catheter ablation procedure (hour 3)
  Rate of acute success at the end of the procedure, i.e. after CT-channels ablation and targeting of the potential remaining VTs, defined as non-inducibility of any VT using a prescribed programmed ventricular stimulation protocol.
Number of VTs persisting at the end of the procedure | end of catheter ablation procedure (hour 3)
  Number of VTs persisting at the end of the procedure
Cycle lengths of VTs persisting at the end of the procedure | end of catheter ablation procedure (hour 3)
  Cycle lengths of VTs persisting at the end of the procedure (ms)
Location of VTs persisting at the end of the procedure | end of catheter ablation procedure (hour 3
  Location of VTs persisting at the end of the procedure with respect to CT channels. Location (critical isthmuses) will be identified using conventional pace mapping or VT/entrainment mapping methods, and described as matching or not matching the location of one CT channel (yes/no/NA)
Rate of VT recurrence at 6-month follow-up | Month 6
  Rate of VT recurrence at 6-month follow-up, defined as at least one appropriate ICD therapy (antitachycardia pacing or shock).
number of sustained VT episodes | Baseline, Month 6
  Efficacy in reducing VT burden, defined as the number of sustained VT episodes detected by the ICD in the 6 months before vs. 6 months after image-guided VT ablation.
Mortality at 6 months follow-up | Month 6
  Mortality at 6 months follow-up
Total procedure duration | end of catheter ablation procedure (hour 3)
  Total procedure duration, defined as the total skin-to-skin time
Procedure duration from start to first radiofrequency ablation | end of catheter ablation procedure (hour 3)
  Procedure duration from start to first radiofrequency ablation
Total radiofrequency ablation time. | end of catheter ablation procedure (hour 3)
  Total radiofrequency ablation time.
Procedure duration from start to completion of CT channels ablation | end of catheter ablation procedure (hour 3)
  Procedure duration from start to completion of CT channels ablation.
Serious adverse effects | Baseline, Month 6
  Major procedure-related complications, including any complication that is potentially life-threatening or that prolongs hospitalization

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Cardiac Pacing and Electrophysiology, CHU Bordeaux, Pessac, France
- Heart Centre, Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided